CLINICAL TRIAL: NCT04028726
Title: Skeletal Muscle Protein Synthesis After Performance of Traditional and Cluster Set Configurations in Resistance-Trained Young Adults
Brief Title: Skeletal Muscle Protein Synthesis: Traditional and Cluster Sets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Texas Christian University (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16987
Record Dates: First submitted 2018-08-02; First posted 2019-07-23 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Resistance Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cluster set Resistance Training Protocol (Active Comparator): Cluster set configuration is the new training approach that it is being tested.
  Interventions: Other: Back-squat exercise
- Traditional Resistance Training Protocol (Sham Comparator): Traditional is commonly used in training sessions.
  Interventions: Other: Back-squat exercise

INTERVENTIONS:
Other: Back-squat exercise — Participants begin with a 5 min dynamic warm-up. Then, they will perform two sets of five repetitions at 40-60% of predetermined 1-repetition maximum (1-RM). The clustered bout will be 4 sets of 2 clusters of 5 repetitions with a 30-second intra-set rest between clusters, and 90-second inter-set rest at a load 70% of 1-RM. The traditional bout will be 4 sets of 10 repetitions with a 120-second inter-set rest at a load 70% of 1-RM.

SUMMARY:
Traditionally, when performing resistance exercise, repetitions are performed in a continuous manner resulting in a decrease in velocity, and thus power output. "Cluster" set is an alternative to counter the reduction in velocity and power output. Cluster sets incorporate a brief rest (15-30 seconds) between individual repetitions (inter-repetition rest) or group of repetitions (intra-set rest) within a set of resistive exercise. In contrast to traditional set configurations, which result in an almost linear decrease in force, velocity, and power -cluster sets maintain and/or attenuate the loss in power, primarily due to higher velocities.

The purpose of this research is to compare the muscle protein synthesis response to acute bouts of cluster and traditional set configurations. Investigators will assess muscle protein synthesis rates before and after acute resistance exercise in 14 resistance-trained males and females (Age: 20-35; back squat 1.5 x body weight; 3 years of resistance training experience). The volunteers are required to be removed (at least six weeks) from all ergogenic levels of nutritional supplements that have previously been shown to affect protein synthesis. Blood and muscle biopsies will be collected as a part of testing. Further, subjects will be required to perform moderate-to-high intensity resistance exercise.

DETAILED DESCRIPTION:
The present study will be testing the effect of rest configuration on muscle protein synthesis. The protocols selected by the researchers were cluster set and traditional set, details will be explained further.

Prior to participation, procedures of the study and the associated risks will be explained to participants prior to enrolling them in the study. Subjects who are interested in participating will be asked to read and sign an informed consent form. If they chose to do so, they will then fill out a medical history questionnaire. Those meeting entry criteria, as identified in the section on Inclusion and Exclusion Criteria, will have their height and weight recorded and blood pressure assessed through use of a blood pressure cuff, followed by determination of body composition by dual x-ray absorptiometry (DXA). DXA is a procedure used to provide researchers with information about body composition using two low dose x-rays. Briefly, participants will be asked to remove all metal objects. They will then be asked to lie on the DXA table where they will be positioned by a trained technician for accurate measurement. The total time of the body composition scan lasts approximately 6-10 minutes depending on the size of the participant. Following determination of body composition, participants will be asked to perform the back squat exercise after demonstration by trained personnel for familiarization with the exercise protocol. The total time associated with consent, body composition assessment, and initial familiarization is approximately 1 to 1.5 hours.

Each participant will be asked to participate in 2 experimental infusion trials, each separated by ≥7 days (Figure 2). The trials will differ in the specific resistance exercise bout performed (CLU or TRD conditions). A standardized evening meal will be provided the night before each experimental infusion. Participants will receive this meal on the 1RM testing day with instructions on when to consume it. Participants will be asked to refrain from any vigorous activities outside of daily living for 72 hours prior to each infusion trial. This will prevent a potential confounding of recently performed exercise on rates of muscle protein synthesis. In addition, subjects will be asked to record their food intake for 3 d before the start of each test day in a food diary that will be provided during the screening.

Subject Activity: On the days of the test, the subject is asked to arrive to Freer Hall by public transport or car in the morning at 8.00 am without eating breakfast (i.e., in the fasting state). After arrival, they will rest on a bed for the majority of the test day (8 - 9.5 h in total). They will perform multiple sets of the back squat exercise with a moderate load (70-75% 1RM) at approximately 10.00 am to 11.00 am each test day. Hereafter, they are asked to rest on a bed again for the remainder of the test day. They will have free access to a restroom, and will be able to work on their laptop, read a book, or watch DVDs during the test day with the exception of during the muscle biopsy procedures.

The resistance training protocols: Participants will perform a dynamic warm-up lasting approximately 5-10 minutes. Following the warm-up, participants will perform two sets of the back squat exercise using a barbell and weight plates with a load equivalent to 40-60% 1RM, as determined through the previous 1RM testing. After 1-2 minutes' rest, participants will perform the back squat using either traditional (4 sets of 10 repetitions with 120 seconds rest) or cluster (4 sets of two clusters of 5 repetitions with 30 seconds between clusters [intra-set rest] and 90 seconds between sets [inter-set rest]) set configurations with a load equivalent to

~70-75% 1RM.Participants will perform both protocols separated by at least 7 days (randomized), thus two trials will be performed. Participants will be asked to perform each repetition as explosively as possible. All testing will be performed on force plate with linear position transducers connected to the bar for determination of force, velocity, and power during the performance of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Resistance-trained adults
* Back squat 1.5x body weight
* 3 years resistance-training experience
* Aged between 20-35 years

Exclusion Criteria:

* Tobacco use (previous 6 months)
* Alcohol consumption >10 drinks per week
* Metabolic disorders, diabetes, thyroid disease, hypogonadism
* Heart disease, arrhythmias, asthma
* History of uncontrolled hypertension
* Orthopaedic injury/surgery within the last year
* Hepatorenal, musculoskeletal, autoimmune, neuromuscular, or neurologic disease
* Consumed ergogenic levels of nutritional supplements that may affect muscle mass (i.e. creatine, HMB), insulin-like substances, or anabolic/catabolic pro-hormones (i.e. DHEA) within six weeks prior to the onset of the study
* Individuals consuming thyroid, androgenic, or other medications known to affect endocrine function
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti- inflammatories, or prescription strength acne medications)
* Pregnant

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Fractional Synthetic Rate of Myofibrillar Proteins | Postabsorptive for 2 hours, Postprandial for 5 hours
  Myofibrillar muscle protein synthesis rates will be assessed during the 2hr Postabsorptive period (e.g. non-fed state) and the 5hr postprandial period (e.g. fed state) for both experimental interventions (e.g. leucine and leucine peptide). This will allow us to assess the change in fractional synthetic rate from the Postabsorptive period to the postprandial period.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Burd, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No